CLINICAL TRIAL: NCT03397290
Title: Usefulness of Bedside Ultrasound in Detection of Pneumothorax Post Transthoracic Lung
Brief Title: Bedside Ultrasound in Detection of Pneumothorax Post Transthoracic Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20170774-01H
Record Dates: First submitted 2017-10-31; First posted 2018-01-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Pneumothorax
Keywords: Chest X-ray; Ultrasound
MeSH Terms: conditions — Pneumothorax | interventions — Ultrasonography; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound Imaging (Experimental): A Single Ultrasound Imaging to diagnose of pneumothorax post transthoracic lung biopsy.
  Interventions: Device: Ultrasound (US) Imaging

INTERVENTIONS:
Device: Ultrasound (US) Imaging — Ultrasound (US) Imaging will be compared to the chest X-ray for diagnostic accuracy (sensitivity and specificity) in diagnoses of pneumothorax post transthoracic lung biopsy

SUMMARY:
Currently chest X-ray (CXR) is the modality used to assess for pneumothorax after transthoracic lung biopsy at the Ottawa Hospital. Recently bedside Ultrasound (US) has become a useful rapid imaging modality to assess chest for pneumothorax in emergency rooms with reported sensitivity, specificity and diagnostic accuracy were 88%, 97% and 97%, respectively (ref. 2).

Our team will be comparing the diagnostic accuracy of US to CXR in diagnoses of pneumothorax post transthoracic lung biopsy.

The purpose of the study is to compare the diagnostic accuracy of US to CXR post-biopsy to confirm the presence of a pneumothorax.

DETAILED DESCRIPTION:
Hypothesis:

US have sensitivity and specificity equal or better than CXR to exclude pneumothorax after transthoracic lung biopsy.

Clinical relevance:

Pneumothorax is a well-known complication of image-guided transthoracic biopsy of lung lesions. The incidence of pneumothorax in patients undergoing TTNB has been reported to be from 9% to 54% (ref. 3). Most of the time, the pneumothorax is small and requires no further intervention other than observation and a repeat CXR to ensure stability or resolution of the pneumothorax. In small group of patients with detected pneumothorax after biopsy, the pneumothorax is either large or becomes larger (more than 2 cm width at the level of the hilum) during observation. In these cases, a small pleural drainage catheter will be inserted to prevent the lung from collapsing. The catheter will be removed in 2 days. Detection of pneumothorax post biopsy is important to prevent possible lung collapse after discharge and currently is done by obtaining a CXR, 30 minutes after the biopsy.

Obtaining a CXR, requires moving the patient on stretcher to the X-ray room, bringing the patient to upright position, patient holds breath. An X-ray technologist obtains the CXR which will be reviewed by a Radiologist when it becomes available on work station. Then the Radiologist revisits the patient and orders the discharge.

Detection of pneumothorax by US is feasible and compare to current practice with CXR, is faster and do not need moving and repositioning the patient, therefore, more convenient. It can be easily performed at the time of clinical assessment prior to discharge.

Study design/ Methodology:

* All patients coming for lung biopsy will be invited to participate in this study. Information about the one additional US at the time of their biopsy and routine CXR will be explained to the patient by either thoracic radiology fellow or staff radiologist.
* For those who agree to participate, informed Consent will be obtained by the same people mentioned above.
* There will be no change in clinical assessment or decision to discharge the patient after biopsy.
* US will be performed by a trained staff radiologist or thoracic fellow.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are booked and coming for image-guided transthoracic biopsy of a lung lesion to the Ottawa Hospital, General Campus, will be consented and those who agree to added US will be included

Exclusion Criteria:

* Other patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | One year
  To determine if the sensitivity and specificity of US is equal or better than routine CXR in diagnosing pneumothorax post lung biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Anne Schwarz, Ph.D., Study Director — Ottawa Hospital Research Institute
Locations (1):
- Hamid Bayanati, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Quick JA, Uhlich RM, Ahmad S, Barnes SL, Coughenour JP. In-flight ultrasound identification of pneumothorax. Emerg Radiol. 2016 Feb;23(1):3-7. doi: 10.1007/s10140-015-1348-z. Epub 2015 Sep 25. PMID 26407979
- [Background] Shostak E, Brylka D, Krepp J, Pua B, Sanders A. Bedside sonography for detection of postprocedure pneumothorax. J Ultrasound Med. 2013 Jun;32(6):1003-9. doi: 10.7863/ultra.32.6.1003. PMID 23716522
- [Background] Boskovic T, Stanic J, Pena-Karan S, Zarogoulidis P, Drevelegas K, Katsikogiannis N, Machairiotis N, Mpakas A, Tsakiridis K, Kesisis G, Tsiouda T, Kougioumtzi I, Arikas S, Zarogoulidis K. Pneumothorax after transthoracic needle biopsy of lung lesions under CT guidance. J Thorac Dis. 2014 Mar;6 Suppl 1(Suppl 1):S99-S107. doi: 10.3978/j.issn.2072-1439.2013.12.08. PMID 24672704